CLINICAL TRIAL: NCT00645424
Title: A Randomized, 12-Week, Open Labeled Study To Evaluate The Efficacy And Safety Of Once Daily Atorvastatin In Diabetes Mellitus Type 2 With Hyperlipidemia
Brief Title: A Study To Evaluate The Safety And Efficacy Of Atorvastatin In Patients With Diabetes And High Cholesterol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2581123
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental)
  Interventions: Drug: atorvastatin
- Arm B (Experimental)
  Interventions: Drug: atorvastatin
- Arm C (Experimental)
  Interventions: Drug: atorvastatin

INTERVENTIONS:
Drug: atorvastatin — Atorvastatin calcium tablets 10 mg orally once daily in the evening for 12 weeks
  Arms: Arm A
Drug: atorvastatin — Atorvastatin calcium tablets 20 mg orally once daily in the evening for 12 weeks
  Arms: Arm B
Drug: atorvastatin — Atorvastatin calcium tablets 40 mg orally once daily in the evening for 12 weeks
  Arms: Arm C

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of atorvastatin for the treatment of Taiwanese patients with diabetes and high cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Adult Taiwanese outpatients with type 2 diabetes mellitus and high cholesterol
* Hemoglobin A1c levels of ≤10%, LDL-C levels of ≥130 mg/dL, and serum triglyceride levels of <400 mg/dL

Exclusion Criteria:

* Type I diabetes mellitus
* Secondary causes of high cholesterol
* Elevated liver enzymes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2003-12; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Percentage change in LDL-C levels from baseline to Week 12 | Week 12
Percentage of subjects with low-density lipoprotein cholesterol (LDL-C) levels of <100 mg/dL (LDL-C responders) at Week 12 | Week 12

SECONDARY OUTCOMES:
Percentage change from baseline in TC, high-density lipoprotein cholesterol, triglycerides, and high sensitivity C-reactive protein at Weeks 4, 8, and 12 | Weeks 4, 8, and 12
Adverse events at Weeks 4, 8, and 12 | Baseline and at Weeks 4, 8, and 12
Clinical laboratory changes at Weeks 4, 8, and 12 | Screening and at Weeks 4, 8, and 12
Vital signs at Weeks 4, 8, and 12 | Screening and at Weeks 4, 8, and 12
Percentage change in LDL-C levels from baseline at Weeks 4 and 8 | Weeks 4 and 8
Percentage of LDL-C responders at Weeks 4 and 8 | Weeks 4 and 8
Percentage of subjects with total cholesterol (TC) levels of <160 mg/dL (TC responders) at Weeks 4, 8, and 12 | Weeks 4, 8, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Taiwan (5):
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Kaohsiung Hsien
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei
  - Pfizer Investigational Site, Taoyuan Hsien

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581123&StudyName=A%20Study%20To%20Evaluate%20The%20Safety%20And%20Efficacy%20Of%20Lipitor%20In%20Patients%20With%20Diabetes%20And%20High%20Cholesterol